CLINICAL TRIAL: NCT01988623
Title: Pivotal Response Treatment for Individuals With Intellectual Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Antonio Hardan, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-25229
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Intellectual Disabilities; Speech Delay; Language Disorder
Keywords: Intellectual Disabilities; Speech Delay; Language Disorder
MeSH Terms: conditions — Intellectual Disability; Language Development Disorders; Language Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pivotal Response Treatment (PRT) (Experimental)
  Interventions: Behavioral: Pivotal Response Treatment (PRT)

INTERVENTIONS:
Behavioral: Pivotal Response Treatment (PRT)

SUMMARY:
The investigators will assess the efficacy of Pivotal Response Treatment (PRT) in the treatment of communication deficits in children with intellectual disabilities. By collecting information about parent and child functioning before and after PRT, The investigators will be able to determine whether the intervention is effective in improving child communication and reducing parent stress.

ELIGIBILITY:
Inclusion Criteria for Individuals with Intellectual Disabilities:

* Participants will have an age range between 2 and 17.11 years of age inclusive
* Male or female
* Diagnosis of an intellectual disability based on the fourth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR), the 10th revision of the International Statistical Classification of Diseases and Related Health Problems (ICD-10), and an expert clinical evaluation
* have historical evidence of significant abnormal developmental milestones as determined by neurological history
* care provider that will reliably bring subject to study visits, and is trustworthy to provide accurate accounts of services provided to the subject

Inclusion Criteria for Individuals with Speech Delay/Language Disorder:

* Participants will have an age range between 2 and 17.11 years of age inclusive
* Male or female
* Diagnosis of a speech delay based on the fourth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR), the 10th revision of the International Statistical Classification of Diseases and Related Health Problems (ICD-10), and an expert clinical evaluation
* Preschool Language scale (PLS) score of at least 1 standard deviations below age level (for children in the age range of 2-6.11)
* care provider that will reliably bring subject to study visits, and is trustworthy to provide accurate accounts of services provided to the subject

Exclusion Criteria:

* medically unstable (such as having unstable seizures)
* primary diagnosis of Autism Spectrum Disorder (ASD) is exclusionary as determined by the investigators

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2012-09-11; Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on the MacArthur-Bates Communication Development Inventory at 6, 12, and 24 weeks | 6, 12 and 24 weeks
Change from Baseline in communication during parent-child and clinician-child interactions at 6, 12, and 24 weeks | 6, 12 and 24 weeks
Change from Baseline on the Social Responsiveness Scale (SRS) at 6, 12, and 24 weeks | 6, 12 and 24 weeks
Change from Baseline on the Clinical Global Impression Scale at 6, 12, and 24 weeks | 6, 12, and 24 weeks

SECONDARY OUTCOMES:
Change from Baseline on the Vineland Adaptive Behavior Scales, Second Edition (VABS-II) at 6, 12, and 24 weeks | 6, 12 and 24 weeks
Change from Baseline on the Parenting Stress Index (PSI) at 6, 12, and 24 weeks | 6, 12, and 24 weeks
Change from Baseline on the Family Empowerment Scale (FES) at 6, 12, and 24 weeks | 6, 12, and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Y. Hardan, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States